CLINICAL TRIAL: NCT04410055
Title: Effects of Dynamic Standing vs. Static Standing on Subjective Fatigue Symptoms
Brief Title: Non-exercise Physical Activity Intervention
Acronym: STAND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Science and Research Centre Koper (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STAND
Record Dates: First submitted 2020-05-23; First posted 2020-06-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Diabete Mellitus; Aging; Cognitive Change
MeSH Terms: conditions — Diabetes Mellitus | interventions — Sitting Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sitting (Active Comparator): Three hours of sitting condition with ad-libitum breaks for toilet use and stretching. During this condition all cognitive, motor and pain scales were monitored.
  Interventions: Behavioral: Sitting
- Static standing (Active Comparator): Four hours of static standing condition with ad-libitum breaks for toilet use and stretching. During this condition all cognitive, motor and pain scales were monitored.
  Interventions: Behavioral: Static standing
- Dynamic standing (Active Comparator): Four hours of dynamic standing condition with ad-libitum breaks for toilet use and stretching. During this condition all cognitive, motor and pain scales were monitored.
  Interventions: Behavioral: Dynamic standing

INTERVENTIONS:
Behavioral: Sitting — We proposed a dynamic standing approach (working while standing accompanied by small periodic stepping movements) as a more tolerable and thereby more applicative lifestyle modification. To evaluate this form on healthy subjects, three different conditions were applied: 3 hours of sitting, static standing and dynamic standing. Both standing conditions were done with height-adjustable table which was developed at the University of Michigan (Ann Arbor, Michigan, USA)
  Other Names: SIT
  Arms: Sitting
Behavioral: Static standing — We proposed a dynamic standing approach (working while standing accompanied by small periodic stepping movements) as a more tolerable and thereby more applicative lifestyle modification. To evaluate this form on healthy subjects, three different conditions were applied: 3 hours of sitting, static standing and dynamic standing. Both standing conditions were done with height-adjustable table which was developed at the University of Michigan (Ann Arbor, Michigan, USA)
  Other Names: STAT
  Arms: Static standing
Behavioral: Dynamic standing — We proposed a dynamic standing approach (working while standing accompanied by small periodic stepping movements) as a more tolerable and thereby more applicative lifestyle modification. To evaluate this form on healthy subjects, three different conditions were applied: 3 hours of sitting, static standing and dynamic standing. Both standing conditions were done with height-adjustable table which was developed at the University of Michigan (Ann Arbor, Michigan, USA)
  Other Names: DYN
  Arms: Dynamic standing

SUMMARY:
Physical inactivity is prevalent in older adults and poses a risk factor for the development of type 2 diabetes. The aim of this pilot study was to examine the effect of non-exercise physical activity using a standing desk on clinical variables in older adults with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* older participants (65+ years) with clinically confirmed type 2 diabetes
* Body mass index above 25 and less than 40 kg/m2

Exclusion Criteria:

* participants unable to perform a short clinical and motor function test battery (sABC test, Mini-BEST)

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-01-08 (Actual); Primary Completion 2022-01-08 (Estimated); Study Completion 2022-01-08 (Estimated)

PRIMARY OUTCOMES:
Oxygen consumption | change in oxygen consumption between all three conditions, which will be measured with a minimum washout period of 3 days
  Oxygen uptake VO2 (ml/min/kg)

SECONDARY OUTCOMES:
Executive control | change in executive control and cognitive switching levels between all three conditions, which will be measured with a minimum washout period of 3 days
  Executive functions measured with Trail Making Test (seconds)
Attention levels | change in attentional levels between all three conditions, which will be measured with a minimum washout period of 3 days
  Measuring attention with Stroop test (seconds)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dempsey PC, Larsen RN, Sethi P, Sacre JW, Straznicky NE, Cohen ND, Cerin E, Lambert GW, Owen N, Kingwell BA, Dunstan DW. Benefits for Type 2 Diabetes of Interrupting Prolonged Sitting With Brief Bouts of Light Walking or Simple Resistance Activities. Diabetes Care. 2016 Jun;39(6):964-72. doi: 10.2337/dc15-2336. Epub 2016 Apr 13. PMID 27208318
- [Background] Wheeler MJ, Green DJ, Ellis KA, Cerin E, Heinonen I, Naylor LH, Larsen R, Wennberg P, Boraxbekk CJ, Lewis J, Eikelis N, Lautenschlager NT, Kingwell BA, Lambert G, Owen N, Dunstan DW. Distinct effects of acute exercise and breaks in sitting on working memory and executive function in older adults: a three-arm, randomised cross-over trial to evaluate the effects of exercise with and without breaks in sitting on cognition. Br J Sports Med. 2020 Jul;54(13):776-781. doi: 10.1136/bjsports-2018-100168. Epub 2019 Apr 29. PMID 31036563
- [Background] Sui W, Smith ST, Fagan MJ, Rollo S, Prapavessis H. The effects of sedentary behaviour interventions on work-related productivity and performance outcomes in real and simulated office work: A systematic review. Appl Ergon. 2019 Feb;75:27-73. doi: 10.1016/j.apergo.2018.09.002. Epub 2018 Sep 18. PMID 30509536
- [Derived] Marusic U, Muller MLTM, Alexander NB, Bohnen NI. Feasibility and behavioral effects of prolonged static and dynamic standing as compared to sitting in older adults with type 2 diabetes mellitus. BMC Geriatr. 2020 Jun 11;20(1):204. doi: 10.1186/s12877-020-01600-0. PMID 32527223